CLINICAL TRIAL: NCT05123131
Title: Isa-RVD Study: Phase II, Multi-centre, Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of the Combination Regimen Isatuximab, Lenalidomide, Bortezomib, and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Isa-RVD Study in Patients With Newly Diagnosed Multiple Myeloma
Acronym: Isa-RVD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Sanofi (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 19-34
Record Dates: First submitted 2021-09-21; First posted 2021-11-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isa-RVD (Experimental): Isatuximab (IV): 10 mg/kg on Days 1, 8, 15, 22, 29 in Cycle 1; from Cycle 2 onwards, it will be given on Days 1, 15, 29.
  Bortezomib (SQ): 1.3 mg/m² on Days 1, 4, 8, 11, 22, 25, 29, and 32. Lenalidomide (PO): 25 mg/day (10 mg/day for patients with creatinine clearance [CrCl] ≥30 to <60 mL/min) from Day 1 to Day 14 and from Day 22 to Day 35 of each cycle.
  Dexamethasone (IV on the days of Isatuximab and PO on other days):
  20 mg/day on Days 1, 2, 4, 5, 8, 9, 11, 12, 15, 16, 22, 23, 25, 26, 29, 30, 32, and 33.
  If patients are ≥75 years old, dexamethasone will be administered on Days 1, 4, 8, 11, 15, 16, 22, 25, 29 and 32.
  Interventions: Drug: Isatuximab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone (IV)

INTERVENTIONS:
Drug: Isatuximab — Isatuximab (IV): 10 mg/kg on Days 1, 8, 15, 22, 29 in Cycle 1; from Cycle 2 onwards, it will be given on Days 1, 15, 29.
Drug: Bortezomib — Bortezomib (SQ): 1.3 mg/m² on Days 1, 4, 8, 11, 22, 25, 29, and 32.
Drug: Lenalidomide — Lenalidomide (PO): 25 mg/day (10 mg/day for patients with creatinine clearance [CrCl] ≥30 to <60 mL/min) from Day 1 to Day 14 and from Day 22 to Day 35 of each cycle.
Drug: Dexamethasone (IV) — Dexamethasone (IV on the days of Isatuximab and PO on other days): 20 mg/day on Days 1, 2, 4, 5, 8, 9, 11, 12, 15, 16, 22, 23, 25, 26, 29, 30, 32, and 33. If patients are ≥75 years old, dexamethasone will be administered on Days 1, 4, 8, 11, 15, 16, 22, 25, 29 and 32.

SUMMARY:
This study aims to evaluate the stringent Complete Response (sCR) rate by the end of two cycles of induction treatment, defined as the proportion of patients who have achieved sCR, according to International Myeloma Working Group (IMWG) criteria, by the end of two cycles of induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed with MM based on standard IMWG criteria and currently requires treatment.
2. Provided voluntary written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
3. Age ≥18 years, ≤75 years, with patients over the age of 70 requiring CI approval.
4. Measurable disease defined as at least one of the following:

   * Serum M protein ≥0.5g/dL (≥5g/L)
   * Urine M protein ≥200 mg/24 hours
   * Serum FLC assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
5. Screening laboratory evaluations within the following parameters:

   * ANC ≥ 1,000 cells/dL (1.0 x 10^9/L) (growth factors cannot be used within 14 days before first study treatment administration)
   * Platelet count ≥75,000 cells/dL (75 x 10^9/L) if <50% BM nucleated cells are plasma cells, ≥30,000 cells/dL (30 x 10^9/L) if ≥50% of BM nucleated cells are plasma cells (without transfusions required during the 3 days prior to the screening haematologic test)
   * Total bilirubin ≤2.0 X ULN (except patients with Gilbert Syndrome, who are eligible if total bilirubin <3.0 mg/dL)
   * AST (SGOT) and ALT (SGPT) ≤3.0 x ULN
   * Haemoglobin ≥8g/dL
   * Calculated CrCl ≥30 mL/min
6. ECOG performance status ≤ 2 (Appendix B).
7. Participant agrees to be registered into the mandatory Risk Management Programme for Lenalidomide and be willing and able to comply with the requirements of this programme.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Participant is considered eligible for ASCT by the treating physician.

Exclusion Criteria:

1. Prior therapy for MM. Participants who received smouldering treatment qualify to participate as long as the prior treatment was not a CD38 therapy.
2. Diagnosed or treated for another malignancy within 3 years prior to enrolment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, or low risk prostate cancer after curative therapy.
3. Central nervous system involvement.
4. Peripheral neuropathy ≥ Grade 3, or Grade 2 with pain on clinical examination during the screening period.
5. Any medical or psychiatric illness that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study.
6. Concurrent uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, Grade 3 thromboembolic event or myocardial infarction within 6 months prior to enrolment.
7. Prior major surgical procedure or radiation therapy within 4 weeks of initiation of study treatment (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of study treatment)
8. Daily requirement for corticosteroids (equivalent to >10 mg/day prednisone for more than 7 days (except for inhalation corticosteroids). Patients may receive corticosteroids for the management of their MM that should not exceed the equivalent of 160mg of dexamethasone in a 2-week period and should be stable for at least 7 days prior to the initiation of study treatment.
9. Concurrent symptomatic amyloidosis or plasma cell leukaemia.
10. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes).
11. Known active infection requiring parenteral or oral anti-infective treatment within 14 days of start of study treatment.
12. Active hepatitis B or hepatitis C viral infection.
13. Pregnant or breastfeeding female or female who intends to become pregnant during the participation in the study. FCBP unwilling to prevent pregnancy by the use of a highly effective method of contraception for ≥4 weeks before the start of study treatment, during treatment (including dose interruptions), and up to 5 months following the last dose of study treatment and/or who are unwilling or unable to be tested for pregnancy before study treatment initiation (2 negative tests), weekly during first month of treatment and then prior each treatment cycle administration or every 2 weeks in case or irregular menstrual cycles up to 5 months following the last dose of study treatment.
14. Male participants who disagree to practice true abstinence or disagree to use highly effective contraception during sexual contact with a pregnant female or FCBP while participating in the study during dose interruptions and at least 5 months following study treatment discontinuation, even if he has undergone a successful vasectomy.

    Note 1: a FCBP is a female who: 1) has achieved menarche at some time point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months). Note 2: True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
15. Receiving any other investigational agents.
16. Hypersensitivity to steroids, or H2 blockers that would prohibit further treatment with these agents.
17. Inability to tolerate thromboprophylaxis.
18. Hypersensitivity (or contraindication) to dexamethasone, sucrose histidine (as base and hydrochloride salt), boron, mannitol, and polysorbate 80, or to any of the components of the study therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Very Good Partial Response (VGPR) or better rate by the end of two cycles of induction treatment | 84 days
  To evaluate the Very Good Partial Response (VGPR) or better rate by the end of two cycles of induction treatment, defined as the proportion of patients who have achieved VGPR, according to International Myeloma Working Group (IMWG) criteria, by the end of two cycles of induction treatment.

SECONDARY OUTCOMES:
To evaluate complete response (CR) and sCR rate following one year and two years of maintenance therapy. | 3.5 years
To evaluate overall response rate and rate of very good partial response (VGPR) or better following one year of maintenance therapy. | 3.5 years
To evaluate time to VGPR or better. | 3.5 years
To assess negative minimal residual disease (MRD) rate following ASCT and after 1 and 2 years of maintenance treatment. | 3.5 years
To evaluate clinical outcomes including time to progression (TTP). | 3.5 years
To evaluate clinical outcomes including progression-free survival (PFS). | 3.5 years
To evaluate clinical outcomes including overall survival (OS). | 3.5 years
To evaluate clinical outcomes including duration of response (DOR). | 3.5 years
To assess the safety of the Isa-RVD treatment regime based on reported adverse events and toxicity. | 3.5 years
To assess the tolerability of the Isa-RVD treatment regime based on reported adverse events and toxicity. | 3.5 years
To evaluate stem cell yield after mobilization. | 90 days

OTHER OUTCOMES:
To evaluate PFS-2 which is defined as time from registration to disease progression or death (from any cause) on next-line therapy. | 3.5 years
To evaluate the clinical efficacy of the Isa-RVD treatment regime in high-risk cytogenetic subgroups (defined as del(1p), gain of 1q, del(17p), t(4;14), t(14;16), t(14;20)) based on treatment response. | 3.5 years
To explore immune modulatory effects of Isa-RVd through immune profiling (NK, T, and B cells) and T-cell receptor sequencing. | 3.5 years
To compare minimal residual disease detection performed by flow cytometry and next generation sequencing. | 3.5 years
To evaluate patient-reported outcomes (PROs) via quality of life instruments through questionnaire completed by patients. | 3.5 years
To evaluate the duration of and time to sCR and time to CR in the subgroup of non-IgG kappa positive patients. | 3.5 years
To evaluate the CR and sCR rate following induction, ASCT and maintenance treatment in the subgroup of non-IgG kappa positive patients. | 3.5 years
To evaluate the immunogenicity of Isatuximab. | 3.5 years
  To be measured using immunoassays.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Peter O'Gorman, Principal Investigator — Mater Misericordiae University Hospital
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- Ireland (4):
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Waterford, Waterford